CLINICAL TRIAL: NCT02574013
Title: The Impact of Use of a Retractor Sponge on Duration of Hospital Stay and Perioperative Complications in Patients With Colorectal Cancer Undergoing Laparoscopic Colorectal Surgery: the SPONGE Trial
Brief Title: Randomized Controlled Trial for Retractor SPONGE Evaluation in Laparoscopic Colorectal Surgery
Acronym: SPONGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, dr. A.B. Smits, MD PhD, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL49877.100.14
Record Dates: First submitted 2015-09-27; First posted 2015-10-12 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Colorectal Cancer; Surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sponge-assisted surgery group (Experimental): Patients offered surgery with use of the retractor sponge
  Interventions: Device: Endoractor®
- Control group (No Intervention): Patients receiving standard care, i.e. surgery in Trendelenburg position

INTERVENTIONS:
Device: Endoractor® — Endoscopic sponge for retraction of small intestine
  Arms: sponge-assisted surgery group

SUMMARY:
To achieve an adequate visual working field during laparoscopic colorectal surgery without disturbance of the small intestine, patients are positioned in Trendelenburg position. This position results in hemodynamic changes which may increase the risk of cardiopulmonary complications and prolonged hospital stay. Recently, an intraoperative retractor sponge was introduced as alternative for the Trendelenburg position during laparoscopic surgery.

DETAILED DESCRIPTION:
Objective: To study the impact of use of an intraoperative retractor sponge on duration of hospital stay and risk of perioperative complications in patients undergoing laparoscopic surgery for colorectal cancer.

Study design: Randomized controlled trial, nested within a prospective cohort according to the 'cohort multiple randomized controlled trial' (cmRCT) design (clinicaltrials.gov NCT02070146).

Study population: Patients with colorectal cancer who undergo laparoscopic sigmoid of rectal resection, and who have given informed consent to be offered experimental interventions within the prospective cohort. Patient who require open surgery or patients with benign colorectal diseases are excluded for this study.

Intervention: Intraoperative use of the retractor sponge versus usual care, i.e. the Trendelenburg position.

Main study parameters/endpoints: The primary endpoint is hospital stay. Secondary objectives are operation time, blood-loss, fluid balance, body temperature, oxygen therapy and postoperative complications.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The study will be conducted according to the cohort multiple Randomized Controlled Trial (cmRCT) design. Within the PLCRC cohort, we will identify all patients who are eligible for the experimental intervention and who have given informed consent to be invited for future experimental interventions. From this sub cohort, we will randomly select a group of patients to whom we will offer surgery with use of the retractor sponge, which they can accept or decline. Eligible patients from the sub cohort who were not randomly selected will undergo standard treatment, i.e. surgery in Trendelenburg position. We do not expect adverse events in patients in the intervention arm.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed distal colon (sigmoid) or rectal cancer,
2. planned for elective laparoscopic colorectal surgery,
3. performance status WHO 0-2
4. broad consent for randomization within ProspectIve data coLlection initiative on ColoRectal Cancer (PLCRC) cohort

Exclusion Criteria:

1. patients planned for open colorectal surgery or emergency colorectal surgery
2. patients with inadequate understanding of the Dutch language in speech and/or writing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Discharge is based on a checklist

SECONDARY OUTCOMES:
Operation time (minutes) | Intraoperative
Blood-loss (ml) | Intraoperative
Fluid balance (L) | Intraoperative
Postoperative body temperature | Baseline
Postoperative oxygen therapy | Baseline
  Number of participants in need for oxygen therapy leaving the recovery room.
Postoperative complications | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Including cardiac, pulmonary, surgical, infectious and thrombovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Anke B Smits, MD PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Derived] Fahim M, Couwenberg A, Verweij ME, Dijksman LM, Verkooijen HM, Smits AB. SPONGE-assisted versus Trendelenburg position surgery in laparoscopic sigmoid and rectal cancer surgery (SPONGE trial): randomized clinical trial. Br J Surg. 2022 Oct 14;109(11):1081-1086. doi: 10.1093/bjs/znac249. PMID 35909251
- [Derived] Couwenberg AM, Burbach MJ, Smits AB, Van Vulpen M, Van Grevenstein WM, Noordzij PG, Verkooijen HM. The impact of retractor SPONGE-assisted laparoscopic surgery on duration of hospital stay and postoperative complications in patients with colorectal cancer (SPONGE trial): study protocol for a randomized controlled trial. Trials. 2016 Mar 10;17(1):132. doi: 10.1186/s13063-016-1256-x. PMID 26964861